CLINICAL TRIAL: NCT05001815
Title: Continuous Subcutaneous Insulin Infusion Versus Multiple Daily Injection in Pregnant Women With Type 2 Diabetes: A Single-center Open Label Randomized Controlled Trial
Brief Title: CSII Versus MDI in Pregnant Women With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021NFM001
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-07

CONDITIONS: Type 2 Diabetes; Pregnancy in Diabetic
Keywords: type 2 diabetes; pregnancy; continuous subcutaneous insulin infusion; multiple daily injection
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pregnancy in Diabetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous subcutaneous insulin infusion (CSII) (Experimental): Patients with indications will receive continuous subcutaneous insulin infusion (CSII) treatment achieved by patch insulin pump devices.
  Interventions: Device: Continuous subcutaneous insulin infusion (CSII)
- Multiple daily insulin injection (MDI) (Active Comparator): Patients with indications will receive traditional multiple daily insulin injection (MDI) treatment.
  Interventions: Device: Multiple daily insulin injection (MDI)

INTERVENTIONS:
Device: Continuous subcutaneous insulin infusion (CSII) — The CSII device used in this study has access to mobile phone, however, without CGM enhanced function
  Arms: Continuous subcutaneous insulin infusion (CSII)
Device: Multiple daily insulin injection (MDI) — Patients with indication will receive MDI treatment with at least one basal insulin injection plus 2 to 3 prandial insulin injection.
  Arms: Multiple daily insulin injection (MDI)

SUMMARY:
The primary objective of the study is to determine if continuous subcutaneous insulin infusion (CSII) can improve glycemic control in women with type 2 diabetes (T2D) who are pregnant.

DETAILED DESCRIPTION:
In women with diabetes, hyperglycemia is associated with increased rates of maternal and fetal adverse outcomes. Mothers are at increased risk of preeclampsia, deterioration of proteinuria and caesarean sections. Infants of mothers with diabetes have increased rates of congenital anomalies, premature delivery, macrosomia, stillbirth and NICU admissions, as well as increased risks of shoulder dystocia, birth injury, hypoglycemia, hyperbilirubinemia, respiratory distress syndrome, asphyxia and death in the neonatal period. Several studies have shown that pregnancy outcomes can be improved along with better glycemic control. Theoretically CSII could achieve better glycemic control due to its flexibility in adjusting both basal rate and bolus insulin infusion. Several randomized controlled studies have compared the ability of CSII with multiple daily injection (MDI) in glycemic control and improvement of pregnancy outcomes in patients with type 1 diabetes (T1D). However, there is a lack of similar studies in women with T2D. We hypothesize that CSII will assist women with T2D achieve better glycemic control during pregnancy compared to MDI users.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 40 years old
2. Patients with confirmed history of T2D or patients who are newly diagnosed with T2D by oral glucose tolerance test (OGTT) during pregnancy (diagnostic criteria refer to ADA 2020 guideline for T2D).
3. Women with singleton pregnancy at 4 to 20 weeks of gestation, whose blood glucose fails to achieved glucose target after adequate lifestyle intervention with or without the prescription of basal insulin (i.e. fasting blood glucose above 5.3 mmol/L, or one hour postprandial blood glucose above 7.8 mmol/L, or two hour postprandial blood glucose above 6.7 mmol/L), and need to start intensive insulin therapy (MDI or insulin pump) according to the evaluation of endocrinologists.
4. Patients who are willing be followed up by the Third Hospital of Peking University in the whole process of pregnancy until 6 weeks of postpartum, and promise that they will provide the results of relative prenatal examinations and perinatal medical records if they are transferred to another hospital for special reasons.
5. Patients who can pass the compliance test and agree to conduct self-monitoring of blood glucose (SMBG) at least 7 times a day during pregnancy.
6. Patients who volunteer to participate the trial and agree to sign informed consent.

Exclusion Criteria:

1. Patients with T1D, special type of diabetes and gestational diabetes.
2. Patients who have received intensive insulin therapy (MDI or insulin pump) or premixed fixed doses of insulin before enrollment in this trial.
3. Patients who refuse to use insulin pump or CGM devices.
4. Patients who are not recommended by obstetrician to continue their pregnancy due to comorbidity and high risk of pregnancy. The comorbidities include but not limited to the following diseases: proliferative retinopathy, chronic kidney disease (eGFR less than 60 ml /min/1.73 with or without heavy proteinuria), known coronary heart disease and cerebrovascular disease, autoimmune disease, other diseases requiring exogenous glucocorticoid or immunosuppressive therapy.
5. Patients who received inpatient psychiatric treatment within 6 months before enrollment or still using psychiatric drugs.
6. Participated in other intervention studies.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) at 24 weeks of gestation | 24 weeks of gestation
  Glycemic control as measured by time in range (TIR) acquired from retrospective continuous glucose monitoring devices (r-CGM) at 24 weeks of gestation among women with type 2 diabetes mellitus.
Time in range (TIR) at 28 weeks of gestation | 28 weeks of gestation
  Glycemic control as measured by time in range (TIR) acquired from retrospective continuous glucose monitoring devices (r-CGM) at 28 weeks of gestation among women with type 2 diabetes mellitus.
Time in range (TIR) at 34 weeks of gestation | 34 weeks of gestation
  Glycemic control as measured by time in range (TIR) acquired from retrospective continuous glucose monitoring devices (r-CGM) at 34 weeks of gestation among women with type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) and glycosylated serum albumin | 24, 28, 34 weeks of gestation and 6 weeks of postpartum
  Glycosylated hemoglobin (HbA1c) and glycosylated serum albumin in meta-late phase of pregnancy.
TIR calculated by patients' SMBG data | At 4 weeks after randomization, and at 24, 28, 34 and 38 weeks of gestation
  TIR calculated by patients' SMBG data at 4 weeks after randomization, and at 24, 28, 34 and 38 weeks of gestation.
TAR and TBR | At 24, 28 and 34 weeks of gestation
  Time above range (TAR) and time below range (TBR) calculated by CGM data at 24, 28 and 34 weeks of gestation.
Blood glucose fluctuation index | At 24, 28 and 34 weeks of gestation
  Mean amplitude of glucose excursion (MAGE), coefficient of variation (CV) and standard deviation (SD) calculated by CGM data recorded at 24, 28 and 34 weeks of gestation.
The AUC of blood glucose within 24 hours before delivery | Within 24 hours before delivery
  The area under curve (AUC) of peripheral blood glucose within 24 hours before delivery: (a) >7.8 mmol/l or 140 mg/dl (b)>6.7 mmol/l or 120 mg/dl (c) <3.5 mmol/L or <63 mg/dl (d) <2.8 mmol/L or <50 mg/dl.
Hypoglycemic events | From randomization, up to 42 weeks of gestation
  (a)Episodes of severe hypoglycemia requiring assistance. (b)Episodes of mild-moderate episodes of hypoglycemia < 3.5mmol/L (mild) and < 2.8 mmol/L (moderate) from patients' SMBG data or from CGM data defined as AUC <3.5 mmol/L or AUC less than or equal to 2.8 mmol/L for 20 minutes duration. (c) Nocturnal hypoglycemia defined as glucose <3.5 (mild) and <2.8 (moderate) by SMBG or CGM between the hours of 23.00-07.00.
Insulin requirements | 4 weeks after randomization, 24, 28, 34 weeks of gestation and 6 weeks of postpartum.
  The total daily insulin dosage at randomization, 4 weeks after randomization, and 24, 28, 34 weeks of gestation as well as 6 weeks of postpartum.
Hypertension during pregnancy | From randomization, up to 42 weeks of gestation
  Hypertension during pregnancy (up to 42 weeks of gestation): Incidence of worsening of chronic hypertension, gestational hypertension, preeclampsia.
Caesarean sections at delivery | At delivery
  Incidence of caesarean section (primary and total)
Gestational weight gain | 24, 28, 34 weeks of gestation and 6 weeks of postpartum
  Gestational weight gain: Absolute and relative weight gain at 24, 28, 34 weeks of gestation and 6 weeks of postpartum comparing to baseline (4-8 weeks of gestation at the time of enrollment)
Maternal hospital stay | From admission to discharge from hospital due to delivery
  Length of hospital stay including admission for delivery and for other obstetric situations during pregnancy.
Infant birthweight | At delivery
  Infant birthweight (at birth): Infant birthweight>90th centile using customized growth curves; infant birthweight<10th centile using customized growth curves; infant birthweight≥4000g or ≤2500g.
Pregnancy loss | From randomization, up to 28 days after delivery
  Including miscarriage, stillbirth and neonatal death (≤28 days of life).
Infant Outcomes (Gestational week of delivery) | At birth
  Infant Outcomes (at birth): The incidence of preterm delivery (<37 weeks and early preterm <34 weeks) and post-term delivery (>42 weeks).
Infant Outcomes (Apgar score) | At birth
  Infant Outcomes (at birth): Apgar score
Infant Outcomes (Up to first 7 days of infants' life) | Up to first 7 days of infants' life
  The incidence of birth injury, shoulder dystocia, neonatal hypoglycemia with intravenous dextrose.
Infant Outcomes (Up to f first 7 days of life) | Up to first 7 days of infants' life
  Incidence of hyperbilirubinemia, respiratory Distress Syndrome (RDS), NICU admission > 24 hours.
The composite endpoint of infants | Up to first 7 days of infants' life
  The combined adverse outcomes of infants including miscarriage, stillbirth and neonatal death; Neonatal birth injury, shoulder dystocia, neonatal hypoglycemia (requiring intravenous glucose infusion), neonatal jaundice, neonatal respiratory distress syndrome (RDS) and more than 24 hours of treatment in NICU.
Questionnaires (WHO-5 physical and mental health index) | At randomization, 34 weeks of gestation and 6 weeks of postpartum
  The score of World health organization (WHO)-5 physical and mental health index acquired from patients.
  The WHO-5 scale (1998 version) was used to measure the patient's quality of life. The scale contains 5 items which initial points is 0-25. The initial points are multiplied by 4 to obtain the percentage points, ranging from 0 to 100，which are used to monitor possible changes in physical and mental health. 0 represents the worst possible quality of life, 100 represents the best possible quality of life, and a difference of 10% indicates significant changes.
Questionnaires (Self-manage behavior scale) | At randomization, 34 weeks of gestation and 6 weeks of postpartum
  The score of Self-manage behavior scale acquired from patients. Diabetes self-care behaviors includes a range of activities (e.g., eating diabetic food, exercising, glucose monitoring and taking medicine), which were evaluated by the Summary of Diabetes Self-Care Activities (SDSCA). SDSCA, compiled by Toobert in 2000, is an 8-likert scale containing 11 items belongs to 6 dimensions, could estimate general diet, special diet, physical activity, glucose monitoring, foot care and medicine compliance of patients with T2DM. The total scores range from 0 to 77, higher score means better diabetes self- care behaviors.
Questionnaires (Self-efficacy scale for diabetes mellitus) | At randomization, 34 weeks of gestation and 6 weeks of postpartum
  The score of self-efficacy scale for diabetes mellitus acquired from patients. Self-Efficacy for Diabetes (SED), a 5-Likert scale including 9 items, is used to measure patients' self-efficacy. The average score is 1-5 points, and the higher the average score, the higher the self-efficacy level of participants. The effectiveness and internal consistency of the Chinese version of SED are reliable, and the load factors of each factor are between 0.579-0.922.
Questionnaires (Self-rated Anxiety Scale, SAS) | At randomization, 34 weeks of gestation and 6 weeks of postpartum
  The score of Self-rated Anxiety Scale (SAS) acquired from patients. Self-Rating Anxiety Scale (SAS) is used to measure the degree of anxiety in patients. There are 20 items in total. The scores are divided into 4 levels, including 5 (items 5, 9, 13, 17, 19) reverse scoring items and 15 positive scoring items. Add the scores of the 20 items to get the rough score, then multiply it by 1.25 and take the integer part to get the standard score. The higher the standard score, the more serious the degree of anxiety.
Questionnaires (Self-rated Depression Scale, SDS) | At randomization, 34 weeks of gestation and 6 weeks of postpartum
  The score of Self-rated Depression Scale (SDS) acquired from patients. The Self-Rating Depression Scale (SDS) is used to measure the degree of depression in patients. There are 20 items in total, including 10 (items 2, 5, 6, 11, 12, 14, 16, 17, 18, and 20) reverse scoring items, and 15 positive scoring items. The depression severity index can be calculated by the cumulative score of each item divided by 80, which could reflect the degree of depression. The index range is 0.25-1.0, and the higher the index, the more severe the degree of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Other researchers can contact the research group for IPD only for academic research, after the ethics committee re-evaluation and determination that the data transmission did not cause privacy disclosure to patients.